CLINICAL TRIAL: NCT06411431
Title: Early Chest Tube Removal After Surgery for Primary Spontaneous Pneumothorax: A Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSP-RCT
Record Dates: First submitted 2024-04-08; First posted 2024-05-13 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-01

CONDITIONS: Primary Spontaneous Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: Surgical intervention and related care will follow current standard practices with the following items representing the randomized arms under investigation:
  * Subjects within the "Early Removal" group will have their chest tube removed on POD#1, within 24 hours from the end of the surgery.
  * Subjects in the "Standard Removal" group will have their chest tube would be removed on POD#2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Early Chest Tube Removal (Experimental): Subjects within the "Early Removal" group will have their chest tube removed on POD#1 within 24 hours from the end of the surgery.
  Interventions: Procedure: Early Chest Tube Removal; Device: Apical Chest Tube
- Standard Chest Tube Removal (Active Comparator): Subjects in the "Standard Removal" group will have their chest tube kept to suction on POD#1 with removal on POD#2.
  Interventions: Procedure: Standard Chest Tube Removal; Device: Apical Chest Tube

INTERVENTIONS:
Procedure: Early Chest Tube Removal — Subjects within the "Early Removal" group will have their chest tube removed if the following criteria are met on the morning of POD#1:
  * ≤1 cm of apical pleural separation and no other areas of pleural separation
  * No air leak
  * No bloody output or concern for bleeding
  * < 400cc of drainage
  Arms: Early Chest Tube Removal
Procedure: Standard Chest Tube Removal — Subjects within the "Standard Removal" group will have their chest tube removal on POD#2 if the following criteria are met on the morning of POD#1:
  * ≤1 cm of apical pleural separation and no other areas of pleural separation
  * No air leak
  * No bloody output or concern for bleeding
  * < 400cc of drainage
  Arms: Standard Chest Tube Removal
Device: Apical Chest Tube — A single apical chest tube will be placed and connected to a suction device at least -20 mmHg suction.

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) with blebectomy/wedge resection plus pleurodesis is the standard of care for recurrent primary spontaneous pneumothorax (PSP) or, in certain instances, after the first episode. The chest tube from surgery is typically kept to suction until post-operative day (POD) 2 to allow for scarring of the lung to the chest to prevent recurrence. However, the scarring process takes place over a period of weeks and is there no data to support POD#2 as the best time to remove the chest tube. Also, shorter chest tube duration can lower length of stay, patient discomfort, and hospital cost.

The goal of this randomized study is to determine if early removal (POD#1) of chest tube after video-assisted thoracoscopic surgery (VATS) with blebectomy/wedge resection plus chemical pleurodesis for primary spontaneous pneumothorax (PSP):

* has no worse 2-year recurrence rate compared to standard removal (POD#2)
* will lower length of stay compared to standard removal
* will result in less complications or re-interventions compared to standard removal

Participants will be asked to join prior to surgery. Following standard-of-care surgery, participants will be screened for randomization. If still eligible, participants will be randomized for early chest tube removal or standard removal. Early Removal will happen within 24 hours after surgery, with Standard Removal happening day 2 after surgery.

Participants will follow-up with the study team for 2 years on the following schedule:

* In clinic with a chest x-ray 2 weeks after surgery
* By phone 3 months after surgery
* In clinic with a chest x-ray 1 year after surgery
* In clinic with a chest x-ray 2 years after surgery

DETAILED DESCRIPTION:
This study will be a multicentered randomized controlled trial. The trial will recruit all adult subjects (>18 years old) with PSP who are undergoing VATS blebectomy/wedge resection with chemical pleurodesis from participating centers. Subjects will be identified by the surgical team when evaluating a subject with PSP for surgery. If screened eligible and not meeting an exclusion criterion, the trial will be discussed with them, and consent will be obtained.

Subjects will undergo VATS with resection of all visible disease or an apical wedge resection if none is found. The use of reinforced or non-reinforced staple loads is left to surgeons' preference. For pleurodesis, choice of chemical agent is at the desecration of the surgeon and common practice but limited to 3 agents (talc, dextrose, or a tetracycline antibiotic). Surgeons can choose to perform a mechanical pleurodesis as they deem appropriate. A single apical chest tube will be placed and connected to a suction device set to at least -20 mmHg of suction. Subjects will then be admitted overnight.

Subjects will be re-evaluated on the morning of POD#1. Those without an air leak, with <400 cc of non-bloody chest tube output, and having a maximum 1cm of apical pleural separation (as determined by the surgeon) will be eligible for randomization to either early or standard removal of their chest tube.

Randomization will occur in a 1:1 manner, stratified by participating center. Subjects within the "Early Removal" group will have their chest tube removed on postoperative day 1 within 24 hours from the end of the surgery with a follow-up chest x-ray within 6 hours from removal in addition to monitoring of symptoms. If the subject remains stable without developing symptoms (new oxygen requirement, shortness of breath, etc.) or increased pleural separation on x-ray, they will be eligible for discharge with appropriate follow-up.

Subjects in the "Standard Removal" group will keep their chest tube to suction until postoperative day 2. The chest tube would be removed on POD#2 with a follow up chest x-ray within 6 hours. If the subject remains stable without developing symptoms (new oxygen requirement, shortness of breath, etc.) or growth of pleural separation on chest x-ray, they would be eligible for discharge.

Subjects will then follow up in clinic within 2 weeks of the operation with a chest x-ray. A 3-month follow-up phone call will be performed. At 1-year post-operative, subjects again will have standard clinic follow up and chest x-ray. Finally, a 2 year follow up phone call and chest x-ray will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing video assisted thoracoscopic surgery with blebectomy/wedge resection and chemical pleurodesis for primary spontaneous pneumothorax
* Adult patients (> 18 years)

Exclusion Criteria:

* Subjects with history of chest radiation or prior ipsilateral chest surgery
* Tuberculosis or other infectious etiology
* Secondary spontaneous pneumothorax (COPD, cancer, cystic fibrosis, connective tissue disease, sarcoidosis, catamenial, etc.)
* Pneumothorax due to trauma
* Hemothorax or hydropneumothorax
* Immunocompromised subjects: neutropenic, leukopenia, or subjects taking immunosuppressive medication such as chemotherapy, transplant medications, steroid (≥5 mg of prednisone or equivalent), etc.
* Interstitial lung disease
* Children (<18)
* Pregnant women
* Adults unable to consent for themselves
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Pneumothorax | 2 years from surgery

SECONDARY OUTCOMES:
Postoperative Length of Stay | End of Surgery to Discharge, up to 90 days
  Postoperative length of stay is defined from the end of the operation until discharge.
Total length of stay | Admission to Discharge, up to 90 days
  Total length of stay is defined as the time from admission until time subject is discharged.
Chest Tube Duration | End of surgery to removal of chest tube, up to 90 days
  From the end of the operation until the removal of the chest tube placed at the initial VATS with pleurodesis.
Complications | 2 years from surgery
  Complications post-surgery such as pleural separation, pleural effusion, hemothorax, etc.
Need for interventions | 2 years from surgery
  Need for additional interventions post-surgery such as thoracentesis, chest tube placement, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Swedish Cancer Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD